CLINICAL TRIAL: NCT03049085
Title: Effect of Preoperative Aspirin in Patients Undergoing Off-pump Coronary Artery Bypass Grafting: A Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Effect of Preoperative Aspirin in Patients Undergoing Off-pump Coronary Artery Bypass Grafting
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medinet Heart Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Preoperative aspirin-OPCAB
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Coronary Artery Disease; Aspirin
Keywords: OPCAB; ASA; Aspirin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin group (Active Comparator): a 75 mg uncoated aspirin is administered 2 hours prior to OPCAB
  Interventions: Drug: Aspirin
- Placebo group (Placebo Comparator): 75 mg Vit. C is administered 2 hours prior OPCAB
  Interventions: Drug: vitamin C

INTERVENTIONS:
Drug: Aspirin — preoperative uncoated 75 mg Aspirin is administered 2 hours prior OPCAB
  Other Names: Acetylsalicylic acid
  Arms: Aspirin group
Drug: vitamin C — preoperative 75 mg Vit. C (Placebo) is administered 2 hours prior OPCAB
  Arms: Placebo group

SUMMARY:
Effect of Preoperative Aspirin in patients undergoing Off-pump Coronary Artery Bypass Grafting. A double-blind, placebo-controlled, randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients undergoing off-pump coronary artery bypass grafting (OPCAB)
* Patients in whom antiplatelet therapy was stopped 5-7 days prior to OPCAB

Exclusion Criteria:

* Patients undergoing on-pump coronary artery bypass grafting
* Patients in whom antiplatelet therapy was not stopped 5-7 days prior to OPCAB
* Intraoperative conversion to on-pump coronary artery bypass grafting
* Patients with inherited blood-clotting disorders
* Patients undergoing other cardiac operations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Myocardial Injury | 6 hours following OPCAB
  Myocardial injury detected by Troponin T (ng/ml)
Myocardial Injury | 12 hours following OPCAB
  Myocardial injury detected by Troponin T (ng/ml)
Myocardial Injury | 24 hours following OPCAB
  Myocardial injury detected by Troponin T (ng/ml)
Myocardial Injury | 72 hours following OPCAB
  Myocardial injury detected by Troponin T (ng/ml)
Inflammation | 6 hours following OPCAB
  Inflammation detected by CRP (mg/l)
Inflammation | 12 hours following OPCAB
  Inflammation detected by CRP (mg/l)
Inflammation | 24 hours following OPCAB
  Inflammation detected by CRP (mg/l)
Inflammation | 72 hours following OPCAB
  Inflammation detected by CRP (mg/l)
Kidney Injury | 6 hours following OPCAB
  Kidney injury detected by creatinine (mg/dl)
Kidney Injury | 12 hours following OPCAB
  Kidney injury detected by creatinine (mg/dl)
Kidney Injury | 24 hours following OPCAB
  Kidney injury detected by creatinine (mg/dl)
Kidney Injury | 72 hours following OPCAB
  Kidney injury detected by creatinine (mg/dl)
All-cause mortality or MACE up to 30 days after surgery | 30 days after surgery
Myocardial Injury | 6 hours following OPCAB
  Myocardial injury detected by CK-MB (U/l)
Myocardial Injury | 12 hours following OPCAB
  Myocardial injury detected by CK-MB (U/l)
Myocardial Injury | 24 hours following OPCAB
  Myocardial injury detected by CK-MB (U/l)
Myocardial Injury | 72 hours following OPCAB
  Myocardial injury detected by CK-MB (U/l)

SECONDARY OUTCOMES:
Postoperative drainage (ml) | 12 hours and 24 hours following OPCAB
Bleeding complication | < 30 days following OPCAB
  reoperation for bleeding, cardiac tamponade
Blood transfusions (units) | < 30 days following OPCAB

CONTACTS AND LOCATIONS:
Locations (1):
- Medinet Heart Centre, Nowa Sól, Lubusz Voivodeship, Poland